CLINICAL TRIAL: NCT01513486
Title: The Effects of Daily Neuromuscular Electrical Stimulation on Muscle Mass During Short-term One-legged Knee Immobilization in Healthy Young Men
Brief Title: Electrical Stimulation During Immobilization
Acronym: ESDIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Assistant Professor, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MEC 11-3-073
Record Dates: First submitted 2012-01-06; First posted 2012-01-20 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Disuse Atrophy; Immobilization; Neuromuscular Electrical Stimulation
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immobilization with NMES (Experimental): Immobilization with daily NMES
  Interventions: Behavioral: immobilization
- Immobilization without NMES (Placebo Comparator): Immobilization without daily NMES
  Interventions: Behavioral: immobilization

INTERVENTIONS:
Behavioral: immobilization

SUMMARY:
In the present study, the effects of 5 days of lower limb immobilization with or without daily neuromuscular electrical stimulation on muscle mass and muscle fiber characteristics will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged from 18-35 years
* 18.5 < BMI < 30 kg/m2

Exclusion Criteria:

* Smoking
* Performing regular resistance training in the previous 6 months
* Hypertension (according to WHO criteria) [46] and/or cardiovascular disease
* Any back/leg/knee/shoulder complaints which may interfere with the use of crutches
* Use of any prescribed medication
* Type 2 diabetes mellitus
* Any family history of thrombosis
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* Myocardial infarction within the last 3 years
* Use of anti-coagulants

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
muscle mass, muscle fiber size | three days before immobilization, and directly after immobilization (day of cast removal; day 6)

SECONDARY OUTCOMES:
muscle strength measured by quadriceps 1-Repetition Maximum by Leg Extension | three days before immobilization, and directly after immobilization (day of cast removal; day 6)

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands